CLINICAL TRIAL: NCT07126002
Title: 16-Week Yoga Improves Bone Density, Metabolism in Elderly Osteoporosis: A Controlled Trial
Brief Title: Yoga Improves Bone Density and Metabolism in Elderly Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025152H
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis
Keywords: Yoga; Bone mineral density; Bone metabolism
MeSH Terms: conditions — Osteoporosis | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participants in the yoga intervention group attended supervised yoga classes twice per week for 16 weeks. Each yoga session lasted approximately 60 minutes and was conducted by certified yoga instructors. Sessions comprised breathing exercises, structured yoga postures, and relaxation. Heart rate was monitored regularly during sessions to maintain appropriate intensity.
  Interventions: Behavioral: Yoga
- control group (No Intervention): Participants in the control group were instructed to maintain their usual activities and not initiate any new structured exercise programs during the study period

INTERVENTIONS:
Behavioral: Yoga — : Participants in this arm received a structured yoga course intervention for a period of 4 months. Sessions were held twice weekly, with each lasting 60 minutes. The curriculum was specifically designed to be gentle, slow-paced, and low-impact, making it suitable for older adults while emphasizing body awareness, mind-body integration, and psychological regulation. The course content included: breathing exercises (e.g., basic abdominal breathing combined with simple movements), asana (posture) practice (e.g., seated chair exercises, standing poses, prone poses, supine poses, and side-lying poses, emphasizing muscle activation, joint flexibility, bodybalance training, and coordination of breath with movement), and meditation and relaxation (e.g.supine rest, moon breath training, and OM chanting). All classes were instructed by experienced yoga teachers certified by the Yoga Alliance.
  Arms: experimental group

SUMMARY:
This study was designed to evaluate the impact of a 16-week yoga program on BMD, bone metabolism markers, and physical fitness in elderly patients with OP.

DETAILED DESCRIPTION:
To assess the effects of a 16-week yoga intervention on bone mineral density (BMD), bone metabolism, and physical fitness in elderly patients with osteoporosis. This randomized controlled trial enrolled 60 adults aged 50 years or older with clinically confirmed osteoporosis. Based on personal preference, participants were assigned to either a yoga group or a control group. The intervention consisted of supervised yoga sessions conducted twice weekly for 16 weeks. The yoga intervention included physical postures, breathing exercises, and meditation/relaxation techniques. Health outcomes were assessed at baseline, mid-intervention (8 weeks), and post-intervention (16 weeks). Primary outcomes included changes in BMD at the lumbar spine and hips. Secondary outcomes comprised serum levels of osteocalcin, procollagen type 1 N-terminal propeptide (P1NP), β-CTX, 25-hydroxyvitamin D, calcium, phosphate, and performance in physical function tests, including grip strength, chair stand, single-leg balance, and timed up-and-go. This randomized controlled trial aims to find out the effect of yoga intervention on bone mineral density (BMD), bone metabolism, and physical fitness in elderly patients with osteoporosis.

ELIGIBILITY:
Inclusion Criteria：

* age ≥50 years;
* diagnosed with osteoporosis using dual-energy X-ray absorptiometry (DXA);
* able to independently perform required assessments;
* voluntary participation in yoga intervention.

Exclusion Criteria:

* secondary osteoporosis;
* severe cardiovascular, cerebrovascular, hepatic, or renal diseases;
* cognitive impairment;
* severe motor dysfunction;
* regular participation in structured exercise programs, such as yoga or resistance training, within the past six months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
bone mineral density | baseline and 4 month
  assessed by dual-energy X-ray absorptiometry (DXA, HOLOGIC Discovery Wi, Bedford, MA, USA), at lumbar spine and bilateral hips. Osteoporosis was diagnosed according to the World Health Organization criteria based on T-scores.

SECONDARY OUTCOMES:
N-MID Osteocalcin | baseline and 4 month
  N-MID osteocalcin is an important biomarker of bone metabolism, mainly reflecting bone formation activity. It is commonly used in clinical practice to evaluate the efficacy of osteoporosis, bone turnover abnormalities, and anti bone resorption therapy
Procollagen 1 N-terminal Propeptide | baseline and 4 month
  Procollagen I N-terminal propeptide (P1NP) is a biomarker that plays an important role in bone metabolism
β-terminal telopeptide of I collagen (β-CTx) | baseline and 4 month
  β-terminal telopeptide of I collagen (β-CTx) has been reported to be a sensitive biochemical marker of bone turnover
25-hydroxyvitamin D | baseline and 4 month
  25 hydroxyvitamin D (25-OH VitD) is the main storage form of vitamin D in the human body and a core indicator for evaluating the nutritional status of vitamin D. It maintains bone health by regulating calcium and phosphorus metabolism
Lower Limb Major Muscle Group Strength (Quadriceps Femoris, HamstringsTriceps Surae, Tibialis Anterior, lliopsoas) | Baseline, 2 Months Post-ntervention, and 4 Months Post-Intervention
  Assesses the strength of major lower limb muscle groups, including the quadricepsfemoris, hamstrings, triceps surae, tibialis anterior, and iliopsoas. Maximum isometric contraction values for both sides are recorded using a MlCROFET2 standardized electronic dynamometer to comprehensively reflect individual lower limb support and gait stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, Beijing Municipality, China